CLINICAL TRIAL: NCT03921333
Title: Double Blind Randomised Placebo Controlled Investigation Into the Effect of Supplementing Plant Extracts on Gut Health, Immunity and Metabolic Disorders in Healthy Adults
Brief Title: The Effect of a Botanical Plant Extract on Gut Health, Immunity and Metabolic Disorders in Healthy Adults
Acronym: GHIMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roehampton (Other)
Responsible Party: Principal Investigator, DR ADELE COSTABILE, Director of the Study, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LSC18/247
Record Dates: First submitted 2019-04-12; First posted 2019-04-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Contraceptives, Oral

STUDY DESIGN:
Intervention Model Description: Dose response study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose plant extract (Active Comparator): 300 mg
  Interventions: Dietary Supplement: Low dose response efficacy of plant extracts
- Middle dose plant extract (Active Comparator): 500 mg
  Interventions: Dietary Supplement: Middle dose response efficacy of plant extracts
- High Dose plant extract (Active Comparator): 700 mg
  Interventions: Dietary Supplement: High Dose response efficacy of plant extracts
- Placebo control (Placebo Comparator): Cellulose microcrystalline
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Low dose response efficacy of plant extracts — 300mg
  Other Names: Low dose
  Arms: Low dose plant extract
Dietary Supplement: Middle dose response efficacy of plant extracts — 500mg
  Other Names: Middle dose
  Arms: Middle dose plant extract
Dietary Supplement: High Dose response efficacy of plant extracts — 700mg
  Other Names: High Dose
  Arms: High Dose plant extract
Dietary Supplement: Placebo — Cellulose microcrystalline
  Other Names: Placebo control
  Arms: Placebo control

SUMMARY:
There is an enormous increase in diabetes mellitus worldwide, especially in developed countries. Ninety percent of diabetes cases worldwide are of Type II diabetes mellitus (T2DM) as a result of greater prevalence of sedentary lifestyle, unhealthy diet and rise of obesity, as well as an increasing number of elderly populations. T2DM can be attributed to relative deficiency of insulin involving insulin resistance, aberrant synthesis of hepatic glucose and progressive deterioration of pancreatic beta-cell functions resulting in chronic hyperglycaemia. A growing amount of evidence has emerged in the last several years linking various nutrients and food sources with a positive management of T2DM. In in vitro studies, various botanical extracts have been found to significantly inhibit the activity of alpha-glucosidase and alpha-amylase. The inhibition of these enzymes' activity is a rational approach in managing glucose level for borderline and T2DM sufferers as inhibition of both alpha-amylase and alpha-glucosidase activity can profoundly reduce post-prandial increase in blood plasma glucose concentration following a mixed carbohydrate intake. Excessive levels of blood plasma glucose and free fatty acids impose a stressful condition for pancreatic beta-cells and other insulin sensitive cells resulting in the local secretion of pro-inflammatory cytokines and chemokines causing a continuous low levels of abnormal inflammation that alter insulin's action. As the body becomes less sensitive to insulin, the resulting insulin resistance leads to further inflammation, with more inflammation causing more insulin resistance, causing blood plasma sugar levels to continuously increase, eventually resulting in T2DM. In in vitro animal models, various compounds of botanical origin have also been shown to possess anti-inflammatory activities which can be beneficial in managing T2DM.

DETAILED DESCRIPTION:
The aim of this human intervention study is to evaluate the impact of a botanical-based extract on gut health, immunity and metabolic disorders in healthy adults.

ELIGIBILITY:
Inclusion criteria

* Females and males, aged 18 years to 65 years
* Body Mass Index (BMI) 27-35 kg/m2
* Not dieting within the last month and not having lost >5% body weight in the previous year
* Not increased physical activity levels in the past 2-4 weeks or intending to modify them during the study
* Understands and is willing, able and likely to comply with all study procedures and restriction including being willing to follow the nutritional advice
* Able to eat most everyday foods
* Habitually consumes three standard meals a day (i.e. breakfast, lunch and dinner)

Exclusion criteria

* Significant health problems (e.g. hypercholesterolaemia, diabetes, GI disorders)
* Taking any medication or supplements known to affect mineral or glucose metabolism within the past month and/or during the study
* Pregnant, planning to become pregnant or breastfeeding
* History of anaphylaxis to food
* Known allergies or intolerance to foods and/or to the study materials (or closely related compounds) or any of their stated ingredients
* BMI <27 kg/m2 or >35 kg/m2
* Volunteers self-reporting currently dieting or having lost >5% body weight in the previous year
* Participants with abnormal eating behaviour
* Participation in another experimental study or receipt of an investigational drug/product within 30 days of the screening visit
* Volunteers who have significantly changed their physical activity in the past 2-4 weeks or who intend to change them during the study
* Participants receiving systemic or local treatment likely to interfere with the evaluation of the study parameters
* Participants on specific food avoidance diets
* Participants who work in appetite or feeding related areas

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Body weight Measurements | Changes from baseline to 4 and 8 week treatment period with plant extracts
  Weight in kilograms
Body mass Index measurements | Changes from baseline to 4 and 8 week treatment period with plant extracts
  kg/m^2
Monitoring Blood pressure changes | Changes from baseline to 4 and 8 week treatment period with plant extracts
  mm/Hg
Microbiota composition | Changes from baseline to 4 and 8 week treatment period with plant extracts
  DNA profiling from faeces (bacteria numbers/g faeces)
Modulation of blood lipids | Changes from baseline to 4 and 8 week treatment period with plant extracts
  Effects on TC, LDL-C, HDL-C and TAG expressed in mmol/L
Changes in insulin | Changes from baseline to 4 and 8 week treatment period with plant extracts
  Effect of insulin levels expressed in mg/dl
Modulation of immune function by plant extracts | Changes from baseline to 4 and 8 week treatment period with plant extracts
  Cytokines analysis on IL6,IL10, IL2 and TNFa expressed in pg/mL

SECONDARY OUTCOMES:
Dietary assessment | Changes from baseline to 4 and 8 week treatment period with plant extracts
  Food Dietary intake analysis via DietPlan 7

CONTACTS AND LOCATIONS:
Overall Officials: Adele Costabile, Dr, Study Director — University of Roehampton; Steve Trangmar, Dr, Study Director — University of Roehampton
Locations (1):
- Health Sciences Research Centre, Life Sciences Department, University of Roehampton, London, UK, United Kingdom